CLINICAL TRIAL: NCT04311866
Title: Comparative Study in the Clinical Efficacy, Satisfaction and Complications While Treating Walking Spica Cast vs Synthetic Pants in the Management of Pediatric Low-energy Femoral Shaft Fracture. Randomized Clinical Trial
Brief Title: Femoral Pediatric Fractures. Walking Spica Cast vs Synthetic Pants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of material for treatment of the patients
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Carlos A Acosta-Olivo, Clinical investigator, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OR19-00002
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Femoral Shaft Fracture; Pediatric ALL
Keywords: femoral pediatric shaft fractures; walking spica cast; synthetic pants
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spica cast (Active Comparator): Standard practice for the management of the femoral shaft fractures.
  Interventions: Device: Spica cast
- Synthetic fabric (Experimental): Offer resistance, durability and low weight to treatment of femoral shaft fractures
  Interventions: Device: Synthetic pants

INTERVENTIONS:
Device: Synthetic pants — The use of synthetic materials is preferred (glass fiber), resistance, durability and low weight makes them optimal. To give some extra strenght to the cast, fiber strips are placed anterior and posterior at the level of the groin, this can facilitate the transportation of the patient avoiding the use of a bar.
  Arms: Synthetic fabric
Device: Spica cast — The use of the spica cast is a standard practice for the management of the femoral shaft fractures, however its use, under some circumstances has been related to a wrong management of the cast, auto-retrieval, patient discomfort, and a difficult situation trying to maintain personal hygiene for the patient.
  Arms: Spica cast

SUMMARY:
Femoral pediatric shaft fractures are a common orthopedic injury. Conservative treatment is still the preferred method by orthopedic surgeons. The walking spica cast is used in patients between 1 year old and 6 years old, in patients with isolated and low-energy fractures. The use of synthetic materials is preferred (fiber glass) for resistance, durability and low weight makes them optimal.

DETAILED DESCRIPTION:
Femoral shaft fractures are the most common orthopedic injury among the femoral fractures in pediatric patients. Approximately 70% of them, are femoral shaft fractures. In the management of this fractures, child abuse has to be discarded, considering age, history, physical examination and radiographic findings.(1) Gross et al suggest that up to 80% of the children that have not yet learned to walk, have been victims of abuse. Moreover, it is important to discard any other condition that could make the child prone to fractures, myelomeningocele, cerebral palsy, osteogenesis imperfecta, non-ossifying fibroma, etc.

Once the diagnosis is made, several variables have to be brought to account, in order to select a treatment method: associated injuries, fracture characteristics, the capability of obtaining an appropriate reduction, familiar situation and costs.

Conservative treatment is still the preferred method by orthopedic surgeons because of its cost and effectivity. Pavlik harness are used in newborns and children up to 6-12 months, it maintains the fracture aligned, it is comfortable and avoids the risk of complications associated to the cast contact with the skin.(1,2) The walking spica cast is used in patients between 1 and 6 years old. Generally this method of treatment is indicated isolated and low-energy fractures.(1) Patients in this group of age with high-energy or comminuted fractures, may require traction prior to the application of the cast. Also, positive Telescope Test may make the patient candidate to traction. In this test, under general anesthesia, a gentile force is applied along the femur, if a 3 or more centimeters shortening is present, the patient has a 20-fold risk of unacceptable shortening.(3) For the application of a cast in femoral fractures, a flexion of 90° in the hip and knee joints is preferred, because this position relaxes the flexor muscles and the hamstrings, besides, it has a lower incidence of loss of reduction and more easy easiness for transportation.(4) in previous studies there has been a loss of reduction 9 times greater in patients immobilized with the knee in less of 50°. The risk of loss of reduction is elevated twice for each centimeter of initial shortening. (1 cm: 12%; 3 cm: 50%)(5) A long cast is applied on the affected extremity, while a gentile traction is maintained and a valgus mold is applied on the fracture site. The remaining part of the cast is applied to the line of the nipples. Caution has to be taken when applying traction to the extremity because the pressure on the popliteus fossa and peroneal nerve. The use of synthetic materials is preferred (glass fiber), resistance, durability and low weight makes them optimal. To give some extra strength to the cast, fiber strips are placed anterior and posterior at the level of the groin, this can facilitate the transportation of the patient avoiding the use of a bar.

A radiographic follow-up during the first 10 days is important because the position of the reduction during the first 7 through 10 days, predicts in a important manner the final result. The cast is retired at 6 - 8 weeks. The rehabilitation therapy is not usually necessary and the parents need to be advised about a residual limp, which can last a few months.

The patient and his family´s life quality has an important role in this kind of injuries. The immediate application of a spica cast substitutes the bed traction prior to the cast application.(4) Multiple adequations have to be made: vehicle safety and transportation, daily supervision, education, home mobility, and hygiene. The home transportation has been identified as the most problematic issue and as a solution to this problem, families have to acquire a wheel chair. (1,4) Hygiene represents a prevalent issue, of minor importance, and parents should be educated about this problem. The position of the cast at 90°-90° may help to solve this issue.

Surprisingly, the need to be absent at work is not the most mentioned problem by parents,. An average of 3 weeks out of work was needed by parents to take care of their child.

Education and learning of the child is vital because of the development and socialization process that takes place during this age. (4) A home tutor works adequately, even though this represents a economic burden to the family.

Activity recovery after retrieval of the cast, such as running and playing starts until 25 days. Physical education should be postponed for one month after retrieval. (4) Surgical treatment is indicated in patients in school age, because of the quality life burden the prolonged immobilization represents. Among those treatments, the options are external fixation, intramedullary flexible nails, and plate fixation.

ELIGIBILITY:
Inclusion Criteria:

* Simple fractures (transverse or short oblique fracture)
* Less than 2 cm of shortening
* Independent walking ability
* Closed fractures
* Isolated shaft fractures
* Low energy
* Written informed consent by the parents

Exclusion Criteria:

* Polytraumatized patients
* Cranial trauma or spinal cord injury
* Articular extension of the fracture
* History of femoral shaft fracture

Ages: 18 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-01-04 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Bone consolidation | 42 days
  Evaluate the bone consolidation during the follow-up, with standard two position x-ray (anteroposterior and lateral) according to Stans classification. When grade 0 represents the absence of indentifiable bone callus; grade 1 primary bone callus with little or no periosteal new bone formation; grade 2 periosteal new bone formation on both sides of bone, and grade 3 represents periosteal new bone formation in three or four sides of the bone

SECONDARY OUTCOMES:
Bone angulation | 42 days
  Evaluate and compare the angulation in all planes (varus, valgus, antecurvature or recurvatum) in two standard x-ray images (anteroposterior and lateral)
Bone shortening | 42 days
  The shortening it was measured in centimeters in two standard X-ray projections, and compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Acosta-Olivo, PhD, Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Hospital Universitario "Dr. José E. González". Universidad Autónoma de Nuevo León, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Flynn JM, Schwend RM. Management of pediatric femoral shaft fractures. J Am Acad Orthop Surg. 2004 Sep-Oct;12(5):347-59. doi: 10.5435/00124635-200409000-00009. PMID 15469229
- [Result] Anglen JO, Choi L. Treatment options in pediatric femoral shaft fractures. J Orthop Trauma. 2005 Nov-Dec;19(10):724-33. doi: 10.1097/01.bot.0000192294.47047.99. PMID 16314721
- [Result] Buehler KC, Thompson JD, Sponseller PD, Black BE, Buckley SL, Griffin PP. A prospective study of early spica casting outcomes in the treatment of femoral shaft fractures in children. J Pediatr Orthop. 1995 Jan-Feb;15(1):30-5. doi: 10.1097/01241398-199501000-00008. PMID 7883924
- [Result] Hughes BF, Sponseller PD, Thompson JD. Pediatric femur fractures: effects of spica cast treatment on family and community. J Pediatr Orthop. 1995 Jul-Aug;15(4):457-60. doi: 10.1097/01241398-199507000-00009. PMID 7560034
- [Result] Illgen R 2nd, Rodgers WB, Hresko MT, Waters PM, Zurakowski D, Kasser JR. Femur fractures in children: treatment with early sitting spica casting. J Pediatr Orthop. 1998 Jul-Aug;18(4):481-7. PMID 9661858
- [Result] Ferguson J, Nicol RO. Early spica treatment of pediatric femoral shaft fractures. J Pediatr Orthop. 2000 Mar-Apr;20(2):189-92. PMID 10739280
- [Result] Epps HR, Molenaar E, O'connor DP. Immediate single-leg spica cast for pediatric femoral diaphysis fractures. J Pediatr Orthop. 2006 Jul-Aug;26(4):491-6. doi: 10.1097/01.bpo.0000217724.08794.e4. PMID 16791068